CLINICAL TRIAL: NCT03880448
Title: Clinical and Microbiological Evaluation of Metronidazole as a Systemic Antimicrobial Adjunct to Periodontal Surgery in the Treatment of Patients With Periodontitis Positive to Porphyromonas Gingivalis
Brief Title: Metronidazole vs Placebo as Adjuncts to Periodontal Surgery for Patients Positive to Porphyromonas Gingivalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Prof. Elena Figuero, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/207
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Periodontitis; Surgery
Keywords: Disease Progression; Microbiota; Periodontitis/surgery; Periodontitis/therapy; Periodontitis/drug effect; Periodontitis/drug therapy; Periodontal diseases/surgery; Periodontal diseases/therapy; Periodontal pocket/drug therapy; Metronidazole/therapeutic use; Metronidazole; Porphyromonas gingivalis; Systemic antimicrobial/periodontal surgery
MeSH Terms: conditions — Periodontitis; Disease Progression; Periodontal Diseases | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects were randomly assigned to the treatment groups in ascending order according to a balanced distribution system through a computer generated random number design table (random block design). Randomization was balanced according to the smoking habit at the initial visit to ensure homogeneity in the treatment groups.
  The method of allocation concealment selected were opaque envelopes. The research coordinator was responsible for the randomization and patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole + periodontal surgery (Experimental): Periodontal surgery + Metronidazole (metronidazole 500mg/8h/7days)
  Interventions: Drug: Metronidazole; Procedure: periodontal surgery
- Placebo + periodontal surgery (Placebo Comparator): Periodontal surgery + Placebo (cornstarch 500mg/8h/7days)
  Interventions: Drug: Placebo; Procedure: periodontal surgery

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 500mg/8h/7days
  Arms: Metronidazole + periodontal surgery
Drug: Placebo — Cornstarch 500mg/8h/7days
  Arms: Placebo + periodontal surgery
Procedure: periodontal surgery — periodontal surgery

SUMMARY:
The objective of this study is to determine whether the use of a systemic antimicrobial (metronidazole) as an adjunct to periodontal surgery provides additional clinical and microbiological beneficial effects compared to periodontal surgery alone plus a placebo, in patients with non treated periodontitis (stage III and IV) positive to Porphyromonas gingivalis.

DETAILED DESCRIPTION:
Design: pilot, randomized, parallel, placebo controlled and triple blind clinical trial.

Sample: Patients with generalized severe chronic periodontitis (stages III and IV) and positive to Porphyromonas gingivalis who potentially need periodontal surgery were recruited from those who attended the postgraduate program in periodontics at the Complutense University in Madrid.

Patients were randomly assigned to the test group (periodontal surgery + metronidazole) or control group (periodontal surgery + placebo).

Study visits:

* Examiner calibration
* Recruitment of patients. Screening. Data collection (clinical and microbiological variables)
* Phase I

  * Non surgical periodontal therapy (2 visits) performed by second year students.
  * Reevaluation at 6 weeks. Data collection (clinical and microbiological variables).

Identification of study participants (patients with probing pocket depth > 5mm in ≥ 2 teeth per sextant or those presenting multiple sites with probing pocket depth ≥ 5mm and bleeding on probing in ≥ one mouth quadrant and positive to Porphyromonas gingivalis.

The need of the surgical procedure was supervised in every case by more than one experienced periodontist (clinical teachers). Finally patients were randomly assigned to their study groups.

* Phase II. Surgical Periodontal Therapy

  * Periodontal surgery sessions performed by second year students. In the last surgery the patient received a recipient containing the pills (metronidazole or placebo according to randomization) and the instructions for use.
  * Suture removal 1 week after the surgery. Data collection 1 week after antibiotic consumption after the last surgery (patient-centered variables on the side effects of antibiotics). Pills recipients were collected in order to evaluate patient compliance. An individual not involved in the study protocol was in charge of doing the data and recipient collection.
* Phase III. Periodontal Maintenance.

  * Maintenance 1(3 months postsurgery). Data collection (clinical and microbiological variables)
  * Maintenance 2 (6 months postsurgery). Data collection (clinical and microbiological variables)
  * Maintenance 3 (9 months postsurgery).
  * Maintenance 4 (12 months postsurgery). Data collection (clinical and microbiological variables)

Security protocol:

Any patient exhibiting worsening in periodontal clinical parameters during the maintenance phase were excluded from the study and inestable sites were re-treated. Inestable sites were considered those exhibiting clinical attachment loss > 2mm between two consecutive visits (Haffajee et al. 1983) after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized severe chronic periodontitis (Armitage 1999) or periodontitis stages III or IV (Papapanou et al., 2018) that may require periodontal surgery.
* Have at least 10 teeth in function, excluding third molars.
* Present sites with pocket probing depth (PPD) ≥ 6mm in ≥ 2 teeth in ≥ one quadrant
* Present radiographic evidence of ≥ 30 % bone loss in ≥ 30% of the dentition
* Detection of Porphyromonas gingivalis in subgingival samples taken at the screening visit as well as in the post-scaling and root planing visit and processed by culture.
* Systemically healthy patients.

Exclusion Criteria:

* Pregnant or lactating women.
* Systemic pathology and/or taking medication that may affect the periodontal situation and/or patients requiring antibiotic prophylaxis.
* Have received systemic antimicrobial treatment 6 months prior to the beginning of the study.
* Have received periodontal treatment 6 months prior to the beginning of the study.
* Patients allergic to metronidazole.
* Patients allergic to cornstarch.
* Patients who refuse to sign the informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) | 6 weeks after scaling and root planing compared to 12 months after the surgery
  Full mouth measurement at 6 sites per tooth with a manual periodontal probe University North Carolina 15 (UNC-15mm)

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Full mouth measurement of the distance in mm from the gingival margin to the bottom of the periodontal pocket at 6 sites per tooth with a manual periodontal probe University North Carolina 15 (UNC-15mm)
Gingival Recession (REC) | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Full mouth measurement of the distance in mm from the cemento-enamel junction to the gingival margin at 6 sites per tooth with a manual periodontal probe University North Carolina 15 (UNC-15mm)
Full mouth plaque score (FMPS) | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Full mouth measurement at 6 sites per tooth of the presence/abscence of dental biofilm (plaque) with a manual periodontal probe University North Carolina 15 (UNC-15mm). Dichotomous evaluation: 0: absence of plaque; 1: presence of plaque)
Full mouth bleeding score (FMBS) | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Full mouth measurement of the bleeding on probing at 6 sites per tooth with a manual periodontal probe University North Carolina 15 (UNC-15mm). Dichotomous evaluation: 0: absence of bleeding on probing; 1: presence of bleeding on probing)
Furcation lesions | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Measurement of the degree of furcation lesions (0,I,II,III) with a Nabers periodontal probe
Clinical attachment level (CAL) | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Full mouth measurement of the distance in mm from cemento-enamel junction to the bottom of the periodontal pocket (REC+PPD) at 6 sites per tooth with a manual periodontal probe University North Carolina 15 (UNC-15mm)
Total Bacterial Counts | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  A microbiological sample is taken with sterilized paper points from the gingival crevicular fluid and the total bacterial counts (expressed in colony forming units/ml) are analyzed by culture.
Percentage of periodontal pathogens | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Determination of the percentage of the following periodontal pathogens:
  * Porphyromonas gingivalis
  * Tannerella forsythia
  * Aggregatibacter actinomycetemcomitans
  * Prevotella intermedia/nigrescens
  * Parvimonas micra
  * Fusobacterium nucleatum
  * Eikenella corrodens
  * Campylobacter rectus
  * Capnocytophaga sp.
  * Eubacterium sp.
Counts of periodontal pathogens | At baseline (before scaling and root planing), 6 weeks after scaling and root planing (Reevaluation Phase I) and during the maintenance Phase III (3, 6 and 12 months after periodontal surgery)
  Determination of the percentage of the following periodontal pathogens:
  * Porphyromonas gingivalis
  * Tannerella forsythia
  * Aggregatibacter actinomycetemcomitans
  * Prevotella intermedia/nigrescens
  * Parvimonas micra
  * Fusobacterium nucleatum
  * Eikenella corrodens
  * Campylobacter rectus
  * Capnocytophaga sp.
  * Eubacterium sp.
Ocurrence of side effects | 1 week after the last surgery + pills intake (placebo or metronidazole)
  The patient was asked if the had experience any adverse effect and a questionnaire was filled in. (Yes/No)
Adverse Effect Description | 1 week after the last surgery + pills intake (placebo or metronidazole)
  The patient was asked to freely describe the adverse effect he had experienced in the case he had.
Degree of affectation of an adverse effect | 1 week after the last surgery + pills intake (placebo or metronidazole)
  The patient was asked to categorize the degree of affectation of the adverse effect (mild, moderate or severe) in case he had experience any.
Patient Compliance | 1 week after the last surgery + pills intake (placebo or metronidazole)
  The patient was asked to bring the recipient with the pills 1 week after the last surgery in order to evaluate how many of them were left and so evaluate their compliance to the prescription dosage. We calculate the percentage of pills the patient takes according to the prescription (1 pill every 8 hours for 7 days - Total of 21 pills)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Study Director — University Complutense Madrid (UCM)
Locations (1):
- Faculty of Dentistry, University Complutense, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No